CLINICAL TRIAL: NCT03530046
Title: A Double-Blind, Randomized Control Trial of Rapidly Infused High Strong Ion Difference Fluid Versus Hartmann's Solution on Acid-Base Status in Sepsis and Septic Shock Patients in the Emergency Department Hospital Pulau Pinang
Brief Title: High Strong Ion Difference Fluid vs Hartmann's Solution on Acid-Base Status in Sepsis
Acronym: HiSIDSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Responsible Party: Principal Investigator, Yeoh Chun Chiat, Principal Investigator, Clinical Research Centre, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ED-HPP-1701
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Septicemic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High SID fluid (Experimental): Group 1: half-normal saline with addition of 75mEq/L sodium bicarbonate
  Interventions: Combination Product: High SID fluid
- Hartmann's solution (Active Comparator): Group 2: Hartmann's Solution
  Interventions: Combination Product: Hartmann's solution

INTERVENTIONS:
Combination Product: High SID fluid — The fluid will be given to the patient at a rate prescribed by the treating physician according to clinical response for a period of 2 hours or up to maximum 30ml/kg fluid is given, whichever is earlier.
  Arms: High SID fluid
Combination Product: Hartmann's solution — The fluid will be given to the patient at a rate prescribed by the treating physician according to clinical response for a period of 2 hours or up to maximum 30ml/kg fluid is given, whichever is earlier.
  Arms: Hartmann's solution

SUMMARY:
This is a research to study primarily the effect of rapidly infused high strong ion difference (SID) fluid vs Hartmann's solution in altering the pH and bicarbonate level of the patient, who is in sepsis with metabolic acidosis. Half of the study population gets high SID fluid, while the other half will get Hartmann's solution.

DETAILED DESCRIPTION:
Balanced fluids are preferred in initial resuscitation of septic patients based on several recent studies.

The Stewart's concept on acid-base balance predicts that high strong ion difference (SID) fluid thus will increase the pH level.

High SID fluid are specially formulated by adding sodium bicarbonate into half saline solution, the resultant fluid contains sodium= 145mmol/L and chloride=70mmol/L (SID= 75) as compared to Hartmann's solution with the SID of 20.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years
* fulfills 2/3 qSOFA criteria
* presumed infection
* a blood pH at presentation ≤ 7.35
* hyperlactatemia (blood lactate level, >2mmol/L )

Exclusion Criteria:

* existing cardiac failure, major cardiac arrhythmia, advanced chronic kidney disease or end stage failure
* known pregnancy
* suspected dengue
* primary diagnosis is related to burn, trauma, or drug overdose
* if more than 500cc of resuscitation fluid was administered before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
pH change | 2 hours
bicarbonate level change | 2 hours
  mmol/L

SECONDARY OUTCOMES:
Lactate level difference | 2 hours
  percentage
Development of pulmonary edema | 48 hours
30 days all-cause mortality | 30 days
Length of stay | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Chunchiat Yeoh, MD, Principal Investigator — Emergency Department, Hospital Pulau Pinang

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2017-01-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT03530046/SAP_002.pdf
  • Study Protocol (2017-01-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT03530046/Prot_003.pdf
  • Informed Consent Form (2017-01-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT03530046/ICF_004.pdf